CLINICAL TRIAL: NCT02273583
Title: Prospective Clinical Trial Evaluating Metronomic Chemotherapy in Patients With High-grade, Operable, Non-metastatic Osteosarcoma of the Extremity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo de Apoio ao Adolescente e a Crianca com Cancer (Other)
Responsible Party: Principal Investigator, Antônio Sérgio Petrilli, MD, PhD, Grupo de Apoio ao Adolescente e a Crianca com Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLATO 2006
Record Dates: First submitted 2014-07-07; First posted 2014-10-24 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: High Grade Osteosarcoma
Keywords: of the extremity
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance therapy (Experimental): 73 weeks of continuous oral low dose chemotherapy with cyclophosphamide (CPM) and methotrexate (MTX) following 31 weeks of MAP.
  Interventions: Drug: continuous oral cyclophosphamide and methotrexate
- Control (No Intervention): 31 weeks of MAP.

INTERVENTIONS:
Drug: continuous oral cyclophosphamide and methotrexate
  Arms: Maintenance therapy

SUMMARY:
Preclinical models show that a daily antiangiogenic regimen at low-dose may be effective against chemotherapy-resistant tumors. The aim of this study is to evaluate the efficacy of maintenance therapy with continuous oral cyclophosphamide and methotrexate in patients with high grade, operable, non-metastatic osteosarcoma (OST) of the extremities. The primary end point is event-free survival (EFS) from randomization.

DETAILED DESCRIPTION:
The study design includes a backbone of 10 weeks of preoperative therapy using MAP (High-dose methotrexate, cisplatin, and doxorubicin). Following surgery, non-metastatic patients were randomized by blocks to complete 31 weeks of MAP or to receive 73 weeks of maintenance therapy following MAP; while metastatic patients received maintenance therapy in combination with MAP since the beginning of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high-grade malignancy osteosarcoma , biopsy-proven , newly diagnosed , previously untreated . Patients with osteosarcoma as a second malignancy should also be eligible .
2. Patients with any primary site , with or without metastases at diagnosis , will be accepted and treated.
3. Patients < 30 years.
4. Patients must have normal body function and adequate renal function defined as serum creatinine < 1.5 x the normal value or creatinine clearance > 60ml/min/1 ,73m2 .
5. Patients must have adequate hepatic function, defined as total bilirubin < 1.5 x normal, aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) < 2.5 x normal.
6. Patients must have adequate cardiac function defined by a shortening fraction > 27 % by echocardiogram or ejection fraction > 47 % by radioisotopic angiogram .
7. If pre- chemotherapy amputation is necessary, the patient is included in the study and eligible to survival analyzes, however the pathological analyze response will be not performed.

   Obtain material for pathological and molecular study is recommended .
8. Whenever possible a central catheter should be placed against the intensity of chemotherapy and need for forced hydration .
9. Patient or legal guardian must sign a consent form which will be explain the type of treatment and procedures that the patient will be submitted .
10. Time > than 4 weeks between biopsy and initiation of treatment - Restaging

Exclusion Criteria:

1. Disease progression ( increase of at least 20% of the extent of the lesion, taking as reference the smallest measurement recorded from the start of treatment, or the appearance of one or more lesions );
2. Any properly documented clinical situation , which at the discretion of the attending physician , patient can not follow with chemotherapy , for safety reasons ;
3. The evaluation of cardiac aspects will be done carefully , so will exclude patients with 20% reduction in the ejection fraction of the left ventricle compared to baseline or with a ventricular ejection fraction < 45 % regardless of baseline;
4. The patient refusal to continue treatment ;
5. Nephrotoxicity , neurotoxicity and ototoxicity grade 4 ;
6. Delay greater than 40 days for the realization of the next treatment cycle , not related to toxicity;
7. Refusal of surgery ; 8 . Variation above 20% of the recommended dose without justification.

Ages: 1 Day to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 738 (Estimated)
Dates: Start 2006-05; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Event-Free Survival | EFS AT 5 YEARS
  AT 5 YEARS

SECONDARY OUTCOMES:
Overall survival | OS AT 5 YEARS
  AT 5 YEARS

CONTACTS AND LOCATIONS:
Locations (1):
- GRAACC- Institute of Pediatric Oncology, São Paulo, São Paulo, Brazil